CLINICAL TRIAL: NCT06500390
Title: Is the Incidence of Temporomandibular Disorder Increased in the Use of Levonorgestrel Intrauterine System
Brief Title: Temporomandibular Disorder in Use of Levonorgestrel Intrauterine System
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: mirena
Record Dates: First submitted 2024-07-08; First posted 2024-07-15 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Levonorgestrel Adverse Reaction; Temporomandibular Joint Disorders; Temporomandibular Disorder
Keywords: Mirena; Levonorgestrel; Intrauterine system; Temporomandibular disorder
MeSH Terms: conditions — Temporomandibular Joint Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group of patients using levonorgestrel intrauterine system (Experimental): The levonorgestrel intrauterine system use patients group consisted of 50 women who had previously a mirena implanted by a gynecologist at least 3 months ago due to menstrual bleeding and pelvic pain.
  Interventions: Diagnostic Test: Examination of temporomandibular joint and masticator muscles
- Control group of healthy patients (Experimental): The control group included 50 randomized health women who had regular menstrual cycles and were not taking any medication.
  Interventions: Diagnostic Test: Examination of temporomandibular joint and masticator muscles

INTERVENTIONS:
Diagnostic Test: Examination of temporomandibular joint and masticator muscles — The TMJ and the masticatory muscles were evaluated by the same clinician. Patients described symptoms such as preauricular pain, limited mouth opening, deviation or deflection during mouth opening, and joint sounds. All patients were assessed using Okeson's Muscle and temporomandibular joint examination and treatment outcome form. This form records (for both TMJ) tenderness and pain in the masseter, temporalis, lateral pterygoid, medial pterygoid, sternocleidomastoid, trapezius, splenius capitis, and digastric muscles, as well as maximum interincisal distance, restriction of laterotrusion and protrusive movements, joint sounds, deviation or deflection during mouth opening, and the visual analogue score (VAS) for pain in the TMJ.

SUMMARY:
The goal of this clinical trial is to investigate the possible role of levonorgestrel intrauterine system use(LIU) in the pathogenesis of temporomandibular joint disorder (TMD). In this clinical trial, levonorgestrel intrauterine system patients (n=30) aged 25-50 and control group patients (n=30) with the same demographics and age range are used. The main questions it aims to answer are:

To compare the frequency of temporomandibular dysfunction in women using the levonorgestrel intrauterine system with the control group of the same demographic and age range.

The levonorgestrel intrauterine system use group consisted of 50 women who had previously a mirena implanted by a gynecologist at least 3 months ago due to menstrual bleeding and pelvic pain.

The control group included 50 randomised healthy women who had regular menstrual cycles and were not taking any medication.

ELIGIBILITY:
Inclusion Criteria:

* Being a woman
* Having used an intrauterine device for at least 3 months
* Being between the ages of 18-50
* Being in American Society of Anesthesiologists-1 and American Society of Anesthesiologists-2 systemic status

Exclusion Criteria:

* Patients with craniofacial syndrome
* Patients with a history of head and neck trauma
* Isolated muscle tenderness or previous surgery on TMJ
* Patients with rheumatological disorders
* Patients with an additional gynecological disease other than endometriosis
* Lack of cooperation with the patient.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 100 (Estimated)
Dates: Start 2024-01-15 (Actual); Primary Completion 2024-04-15 (Actual); Study Completion 2024-12-15 (Estimated)

PRIMARY OUTCOMES:
Evaluation of temporomandibular joint disorder and masticator muscle pain | One Day
  To measure whether there is any difference in the incidence of temporomandibular joint disorders and masticator muscle pain between two groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Marmara University, Istanbul, Maltepe, Turkey (Türkiye)

REFERENCES:
- [Derived] Can S, Can SBK, Karakus SS, Berkel G. Does the use of the levonorgestrel intrauterine system increase the prevalence of masticatory muscles tenderness? Oral Surg Oral Med Oral Pathol Oral Radiol. 2025 Oct;140(4):384-390. doi: 10.1016/j.oooo.2025.03.001. Epub 2025 Mar 8. PMID 40393879